CLINICAL TRIAL: NCT04864756
Title: Medical Simulation Teaching and Academic Performance Among Medical Students at a Medical School in Rural Uganda
Brief Title: Simulation Based Learning and Academic Performance in Medical School
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other); Alberta Children's Hospital Research Institute (Other); The ELMA Foundation (Other); Laerdal Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/MUST/SIM-II
Record Dates: First submitted 2021-04-17; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Academic Performance

STUDY DESIGN:
Intervention Model Description: Before and after comparison
Masking Description: No masking applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before/After (Experimental): Grade performance before and after introduction of simulation based learning
  Interventions: Other: Simulation based learning

INTERVENTIONS:
Other: Simulation based learning — Learning for medical students using simulation based techniques including scenario execution as a complement to conventional teaching methodologies

SUMMARY:
The investigators will use a multi-methods approach, including both qualitative and quantitative methods. In the quantitative methodology, the investigators will use a before and after approach to compare medical student grades/scores before and after the integration of Simulation based learning (SBL) in the curriculum. The hypothesis is that SBL will generally increase knowledge and skills and hence improve the scores from the theory (MCQ) and clinical (OSCE) examinations conducted outside simulated settings in the clinical departments.

DETAILED DESCRIPTION:
Simulation faculty development will be measured by retention and engagement in simulation sessions. The investigators will use survival analysis methods and plot Kaplan Meier curves to calculate probability of retention and determine the factors that are associated with retention as derived from participant in-depth interviews and departmental meetings. A faculty member will be considered disengaged if they do not participate in simulation session for at least 6 months post training, despite reminders and opportunities for participation. Reasons for potential disengagement will be explored qualitatively.

In the qualitative approach, the investigators will conduct in-depth key informant interviews (45 minutes to 1 hour) with administrators at the institution, namely Academic Registrar, Deans of Medical School, heads of Departments and Simulation facilitators (the post-graduate student trainers). The investigators will conduct focus group discussions (1 hour) with postgraduate simulation facilitators, the medical and nursing students before, during and after their enrollment in SBL. The interviews and focus group discussions will be audio-recorded and transcribed.

ELIGIBILITY:
Inclusion Criteria:

* Medical (Medicine and Nursing) students
* Enrolled in the Faculty of medicine at Mbarara University of Science and Technology
* Currently attending clinical years

Exclusion Criteria:

* Non clinical student years in the Faculty of Medicine
* not enrolled in Medicine or Nursing programs at Mbarara University of Science and Technology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Academic performance | 36 months after introduction of simulation based techniques
  Change in CGPA scores Before and after introduction of simulation based techniques

SECONDARY OUTCOMES:
Retention of academic faculty | 2 years after initiation of simulation based learning
  Percentage of faculty retained in the training program

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data will share with permission from the research ethics committee and Mbarara University Academic Registrar's authorization
Supporting Information: Study Protocol, ICF